CLINICAL TRIAL: NCT04857866
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Study of the Safety, Tolerability, and Pharmacokinetics of XmAb®27564 in Healthy Volunteers
Brief Title: Safety, Tolerability and PK of a Single Subcutaneous Injection of XmAb27564 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XmAb27564-01
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Safety in Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose - XmAb27564 Subcutaneous injection of Dose A, B, C, D, E or F (Experimental)
  Interventions: Drug: XmAb27564
- Single Ascending Dose - Placebo Subcutaneous injection of placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XmAb27564 — Single ascending dose of XmAb27564
  Arms: Single Ascending Dose - XmAb27564 Subcutaneous injection of Dose A, B, C, D, E or F
Drug: Placebo — Single dose of placebo
  Arms: Single Ascending Dose - Placebo Subcutaneous injection of placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending-dose study of subcutaneously administered XmAb27564 or placebo in healthy male and female subjects.

DETAILED DESCRIPTION:
This study will determine the safety and tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of XmAb27564 in normal healthy volunteers. XmAb27564 is an engineered IL-2 mutein being developed for autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Total body weight 50.0 to 100.0 kg and body mass index (BMI) 19.0 to 35.0 kg/m2
* In good general health with no clinically significant abnormality identified on medical or laboratory evaluation and no history of any clinically significant disorder, condition, or disease.
* A nonsmoker for at least 12 weeks preceding screening
* Female subjects of childbearing potential must agree to use a highly effective method of birth control during and for 45 days after administration of investigational product (IP).
* Fertile male and female subjects must be willing to practice a highly effective method of birth control during and for 45 days after administration of IP and agree not to donate sperm from screening through 45 days after administration of IP.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of diseases or disorders that would pose a significant risk to subject's safety or significantly interfere with the study evaluation, procedures, or completion
* Subjects with history of any cardiovascular event
* Subjects with vital sign values outside the normal ranges
* Subjects who are positive for MTB QuantiFERON, hepatitis B surface antigen, hepatitis C virus antibody, severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) by polymerase chain reaction (PCR)/antigen, or human immunodeficiency virus Type I or Type II tests at screening
* Subjects with signs or symptoms consistent with active viral infection
* Subjects with baseline eosinophil elevation or a history of urticaria, asthma, allergic dermatitis, food allergy or eosinophilic esophagitis
* Subjects who have evidence of any bacterial, viral, parasitic, or systemic fungal infections requiring treatment within the 21 days prior to randomization; or hospitalization due to infection within 3 months prior to randomization
* Subjects who have had any prior investigational treatment with interleukin 2 (IL-2) therapies or have received any investigational agent within five half-lives of the study drug
* Subjects with a known or suspected sensitivity to products from mammalian cell lines
* Subjects who have received live vaccines ≤ 2 months prior to screening or any vaccine within the past 14 days

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events, graded by CTCAE Version 5.0 | Up to Day 45

SECONDARY OUTCOMES:
PK: Area Under the Drug Concentration - Time Curve from Zero to the End of Observation | 45 Days
PK: Maximum Observed Drug Concentration (Cmax) of XmAb27564 after a single dose | 45 Days
PK: Measurement of Cmax | 45 Days
PK: Time to Maximum Plasma Concentration (Tmax) of XmAb27564 after a single dose | 45 Days
PK: Measurement of Tmax | 45 Days
PK: Time to Decrease in Concentration by Half (T1/2) of XmAb27564 after a single dose, due to elimination | 45 Days
PK: Measurement of T1/2 | 45 Days
PD: Measurement of Change in Number of Regulatory T Cells | 45 Days
PD: Measurement of Change in Number of Subsets of Conventional T Cells in Blood | 45 Days
PD: Measurement of Change in Number of Natural Killer Cells (NK Cells) in Blood | 45 Days
PD: Measurement of Cytokines in Blood | 45 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zitnik, MD, Study Director — Executive Medical Director, Clinical Development, Xencor
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States